CLINICAL TRIAL: NCT07389694
Title: Modulating Bilateral Cortical Activation In Adults Who Stutter: A Pilot Study
Brief Title: Using Transcranial Magnetic Stimulation to Treat Stuttering
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Responsible Party: Principal Investigator, Kristin Pelczarski, Associate Professor, Kansas State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KPelczarski
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Stuttering, Adult
Keywords: stuttering; noninvasive treatment; transcranial magnetic stimulation; eye tracking; EEG
MeSH Terms: conditions — Stuttering | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Repeated measures, single subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Transcranial Magnetic Stimulation to treat stuttering (Experimental): There is only one arm to this study. All participants will receive 10 days of Transcranial Magnetic Stimulation to specific cortical speech and motor areas.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — This study uses Transcranial Magnetic Stimulation (TMS) applied to specific speech and motor areas of the brain to stimulate cortical areas that experience reduced activations during left-hemisphere dominant tasks in people who stutter.

SUMMARY:
The goal of this clinical trial is to learn if repeated transcranial magnetic stimuli (rTMS) can treat stuttering in adults. The main questions it aims to answer are:

* Will there be changes in the brains of people who stutter because of the treatment?
* Will any changes in the brain result in less stuttering?

Participants will:

* Visit the lab 3 times before treatment for tests
* Complete 10 rTMS sessions
* Visit the lab 2 times after treatment for tests

DETAILED DESCRIPTION:
Measures must be obtained to in preparation for TMS treatment. Structural MRI and resting-state functional MRI (rsfMRI) recordings will be obtained from the participant, and they will undergo a neuronavigational session to determine best placement for the electrodes.

MRI/rsfMRI recordings: The structural MRIs will be obtained and used for TMS neuronavigation. Resting-state functional MRI will be recorded for 8 min with the eyes open. rTMS will be delivered at 10 Hz for 10 min with a stimulation intensity of 120% of the resting motor threshold (rMT).

Neuronavigation: The TMS coil will be navigated with a neuronavigation system using the individual MRIs. rTMS targets: rTMS will be delivered to the left inferior frontal gyrus (IFG). We will use the neuronavigation system to identify the IFG.

Three pre-treatment and 2 post-treatment sessions will each obtain data from the following measurements:

* rs-EEG: rs-EEG responses will be recorded with eyes open for 5 minutes using a 64-channel EEG system.
* Eye tracker: eye gaze fixations, dwell time, saccades, and gaze durations will be recorded while the participant completes several behavioral phonological memory tasks.
* Spontaneous speech sample will be obtained to determine percent syllables stuttered.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years
* Self-identifies as a person who currently stutters
* Right-handed or left-handed
* Normal hearing and (corrected) vision
* Able to understand and give informed consent
* Monolingual English speaker

Exclusion Criteria:

* Cardiac pacemaker or pacemaker wires; neurostimulators; implanted pumps
* Metal in the body (rods, plates, screws, shrapnel, dentures, IUD) or metallic particles in the eye
* Facial tattoos
* Not having medical insurance
* Surgical clips in the head or previous neurosurgery
* Any magnetic particles in the body
* Cochlear implants
* Prosthetic heart valves
* Epilepsy or any other type of seizure history
* History of significant head trauma (i.e., extended loss of consciousness, neurological sequelae)
* Known structural brain lesions
* Pre-existing speech, language, or neurological disorder (except for stuttering)
* Significant other disease (heart disease, malignant tumors, mental disorders)
* Significant claustrophobia; Ménière's disease
* Women who are trying to get pregnant and sexually active women (of reproductive age) not on a reliable contraceptive
* Pregnancy, breastfeeding
* Medications increasing the risk for seizures
* Non-prescribed drug use
* Use of recreational drugs such as medical marijuana
* Failure to perform the behavioral tasks or neuropsychological evaluation tests
* Prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Changes in functional connectivity with resting-state electroencephalography (rs-EEG) | Baseline, immediately post-treatment, and one week after post-treatment.
  A seed-based functional connectivity analysis will be carried out between the two stimulated brain areas. To assess the changes in effective connectivity, the investigators will compare the seed-based connectivity values across sessions.
Changes in behavioral measures of stuttering and phonological processing. | Baseline, immediately post-treatment, and one week after post-treatment.
  To assess functional changes as a result of rTMS treatment, comparison of eye tracking measurements of duration, dwell time, and number of fixations of eye movements while completing speech and language-based tasks are compared across sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Pelczarski, Ph.D., Principal Investigator — Kansas State University; Julio Hernandez Pavon, Ph.D., DSc, Principal Investigator — Kansas State University
Locations (1):
- Bluemont Hall, Department of Psychological Sciences, Kansas State University, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication with be shared with other researchers.

REFERENCES:
- [Background] Ridding MC, Rothwell JC. Is there a future for therapeutic use of transcranial magnetic stimulation? Nat Rev Neurosci. 2007 Jul;8(7):559-67. doi: 10.1038/nrn2169. PMID 17565358
- [Background] Hernandez-Pavon JC, Harvey RL. Noninvasive Transcranial Magnetic Brain Stimulation in Stroke. Phys Med Rehabil Clin N Am. 2019 May;30(2):319-335. doi: 10.1016/j.pmr.2018.12.010. Epub 2019 Feb 21. PMID 30954150
- [Background] Hernandez-Pavon JC, Veniero D, Bergmann TO, Belardinelli P, Bortoletto M, Casarotto S, Casula EP, Farzan F, Fecchio M, Julkunen P, Kallioniemi E, Lioumis P, Metsomaa J, Miniussi C, Mutanen TP, Rocchi L, Rogasch NC, Shafi MM, Siebner HR, Thut G, Zrenner C, Ziemann U, Ilmoniemi RJ. TMS combined with EEG: Recommendations and open issues for data collection and analysis. Brain Stimul. 2023 Mar-Apr;16(2):567-593. doi: 10.1016/j.brs.2023.02.009. Epub 2023 Feb 23. PMID 36828303
- [Background] Pelczarski KM, Tendera A, Dye M, Loucks TM. Delayed Phonological Encoding in Stuttering: Evidence from Eye Tracking. Lang Speech. 2019 Sep;62(3):475-493. doi: 10.1177/0023830918785203. Epub 2018 Jul 6. PMID 29976115
- [Background] Pelczarski KM, Yaruss JS. Phonological memory in young children who stutter. J Commun Disord. 2016 Jul-Aug;62:54-66. doi: 10.1016/j.jcomdis.2016.05.006. Epub 2016 May 17. PMID 27280891
- [Background] Pelczarski KM, Yaruss JS. Phonological encoding of young children who stutter. J Fluency Disord. 2014 Mar;39:12-24. doi: 10.1016/j.jfludis.2013.10.003. Epub 2013 Nov 20. PMID 24759190
- [Background] Byrd CT, McGill M, Usler E. Nonword repetition and phoneme elision in adults who do and do not stutter: Vocal versus nonvocal performance differences. J Fluency Disord. 2015 Jun;44:17-31. doi: 10.1016/j.jfludis.2015.01.004. Epub 2015 Jan 24. PMID 25680736
- [Background] Anderson JD, Wagovich SA, Hall NE. Nonword repetition skills in young children who do and do not stutter. J Fluency Disord. 2006;31(3):177-99. doi: 10.1016/j.jfludis.2006.05.001. Epub 2006 Jun 30. PMID 16814376
- [Background] Strand F, Forssberg H, Klingberg T, Norrelgen F. Phonological working memory with auditory presentation of pseudo-words -- an event related fMRI Study. Brain Res. 2008 May 30;1212:48-54. doi: 10.1016/j.brainres.2008.02.097. Epub 2008 Mar 18. PMID 18442810
- [Background] Perrachione TK, Ghosh SS, Ostrovskaya I, Gabrieli JDE, Kovelman I. Phonological Working Memory for Words and Nonwords in Cerebral Cortex. J Speech Lang Hear Res. 2017 Jul 12;60(7):1959-1979. doi: 10.1044/2017_JSLHR-L-15-0446. PMID 28631005
- [Background] Neef NE, Anwander A, Butfering C, Schmidt-Samoa C, Friederici AD, Paulus W, Sommer M. Structural connectivity of right frontal hyperactive areas scales with stuttering severity. Brain. 2018 Jan 1;141(1):191-204. doi: 10.1093/brain/awx316. PMID 29228195
- [Background] Neef NE, Hoang TN, Neef A, Paulus W, Sommer M. Speech dynamics are coded in the left motor cortex in fluent speakers but not in adults who stutter. Brain. 2015 Mar;138(Pt 3):712-25. doi: 10.1093/brain/awu390. Epub 2015 Jan 15. PMID 25595146